CLINICAL TRIAL: NCT02280330
Title: Iodine Intake & Status of Preschoolers Given Micronutrient Powder for 6 Months
Brief Title: Iodine Status of Preschoolers Given Micronutrient Powder for 6 Months
Acronym: MNP-CAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nutrition Center of the Philippines (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NCP-RPU-2014-0001
Record Dates: First submitted 2014-10-27; First posted 2014-10-31 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Iodine Deficiency; Iodine Deficiency Disorder; Hypothyroidism
Keywords: Iodine Deficiency; Micronutrient Powder; Hypothyroidism
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MNP group (Active Comparator): The MNP group will receive 60 sachets of MNP in a period of 6 months or 10 sachets per month equivalent to 3-4 sachets in a week.
  Interventions: Dietary Supplement: MNP group
- Placebo group (Placebo Comparator): The placebo group will receive 60 sachets of placebo (with same characteristics) as the MNP or 10 sachets per month equivalent to 3-4 sachets in a week.
  Interventions: Other: Placebo group

INTERVENTIONS:
Dietary Supplement: MNP group — MNP contains 15 vitamins an minerals, including Vitamin ADEC, B1, B2, B6, B12, Niacin, Folic Acid, Iron, Zine, Copper, Selenium and Iodine. There is 90 microgram of iodine per sachet of one gram of MNP.
  Other Names: Multinutrient Powder
  Arms: MNP group
Other: Placebo group — The placebo is maltodextrin which is prepared as a white powder with similar physical characteristics and taste as MNP.
  Other Names: Placebo
  Arms: Placebo group

SUMMARY:
Iodine deficiency remains widespread worldwide with children as among the vulnerable groups considering their stage of growth and development. In the Philippines, current data shows an optimal status among schoolchildren, however no data exists on iodine status nor intake of preschool children. One recent approach to improvement of the vitamin and mineral status of the population is home fortification using micronutrient powder or MNP. This contains 15 vitamins and minerals, including iodine and iron. Current guidelines exist for MNP use to improve iron status and reduce anemia among infants and young children 6-23 months old, but did not mention use among preschoolers such as those in day care centers. This study, therefore, aims to compare the iodine status and growth of day care children given MNP for 6 months.

DETAILED DESCRIPTION:
Iodine is an essential trace element for normal growth and development in animals and man (Hetzel, 1989). When iodine requirements are not met, thyroid hormone synthesis is impaired resulting in hypothyroidism and a series of functional and development abnormalities called iodine deficiency disorders or IDD develop (WHO, 2007).

WHO estimated that two billion people worldwide, including 1/3 of school-age children (de Benoist et al. cited by Zimmerman, 2011) suffer from iodine deficiency. Evidence is lacking as to whether schoolchildren are good proxy for other groups such as young children (Sullivam, 2010). In the Philippines, no data exists on the iodine status of preschool children.

One recent approach for improving the vitamin and mineral status of the population is the use of micronutrient powder which contains 15 vitamins and minerals including iodine (HF-TAG 2011). While the MNP has been found effective to improve iron status, its effectiveness in improving iodine status has yet to be studied. Further, the provision of iodine through MNPs as well as the combined impact of salt iodization and use of MNPs, warrant investigation. It would also be of interest to generate data on the knowledge, attitude and practices of their parents or other caregiver who primarily take care of planning and provision of food for the family on iodine, iodized salt and MNP.

Day care centers (DCC) are chosen as the site of the study considering their conduct of 120-days supplementary feeding yearly and the organized structure presents a better compliance and easier monitoring of use. Further, the day care pupils, more or less, represent the preschoolers in the barangay and there may be commonality (homogeneity) of the children in age and other characteristics.

In the absence of guidelines for MNP use among children 24 months or older, the existing guidelines such as 60 sachets in 6 months as stipulated in DOH AO 2011-0303 will be followed.

ELIGIBILITY:
Inclusion Criteria:

* apparently healthy
* permanent resident in the barangay or municipality
* 4-6 years old
* with informed written parental consent
* whose mothers are willing to devote time for the survey

Exclusion Criteria:

* severely underweight
* with obvious clinical problem like goiter, congenital heart disease
* with plans of transferring residence outside the municipality within the next 6 months

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 396 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Iodine status based on urinary iodine measures | 6 months

SECONDARY OUTCOMES:
Change in growth as indicated by anthropometric parameters such as weight for age and height for age | 6 months
Levels of iodine intake | 6 months
Association of child characteristics with iodine intake | 6 months
  Child characteristics include age, birth order, common illnesses
Association of mother/caregiver characteristics with iodine intake | 6 months
  Mother / Caregiver information includes age, religion, ethnic tribe, educational attainment, occupation and economic role in the family
Association of household characteristics with iodine intake | 6 months
  Household information includes status of residence, length of residence, type of residence, nature of living arrangement, source of drinking water, household number, main source of income and estimated family income
Association of environmental sanitation with iodine intake | 6 months
  Environmental sanitation includes garbage disposal, drinking water, house premise, handwashing
Likability of a communication material on the knowledge of the mothers/caregivers regarding iodine, iodized salt and micronutrient powder | 6 months
  Included here is a survey on preference of communication material, preferred size, color and topic for Iodine, Iodized salt and micronutrient powder

CONTACTS AND LOCATIONS:
Overall Officials: Imelda O Degay, Principal Investigator — University of the Philippines Los Banos
Locations (1):
- La Trinidad Benguet Day Care Centers, La Trinidad, Benguet, Philippines